CLINICAL TRIAL: NCT04461730
Title: Role of Basal Ganglia and Thalamus in Perceptual Consciousness and Metacognition
Acronym: METACTION
Status: Withdrawn | Type: Observational
Why Stopped: team no more available to lead research
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.271; 2019-A02328-49 (Other: ID RCB)
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease; OCD; Dystonia
Keywords: metacognition; consciousness; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Parkinson disease
  Interventions: Device: deep brain stimulation
- essential tremor
  Interventions: Device: deep brain stimulation
- dystonia
  Interventions: Device: deep brain stimulation
- OCD
  Interventions: Device: deep brain stimulation
- healthy volunteers

INTERVENTIONS:
Device: deep brain stimulation — Behavioral and electroencephalographic responses will be compared on and off deep brain stimulation
  Groups: OCD; Parkinson disease; dystonia; essential tremor

SUMMARY:
The term perceptual awareness refers to subjective experience... or the phenomenology associated with the processing of a sensory stimulus. The term metacognition refers to our ability of introspection, knowledge and control of our own cognitive processes. The objective of this research is to establish the contribution of the basal ganglia and thalamus to the perceptual awareness and meta-cognition, using deep brain stimulation coupled with electroencephalography.

ELIGIBILITY:
Inclusion Criteria:

* Major patient in need of brain stimulation therapy for motor disorders (Parkinson's disease, tremor, dystonia) or psychiatric disorders (OCD).
* Outpatient or inpatient follow-up
* Fluent in French and able to understand the study procedures
* informed consent
* Patient affiliated to social security
* Written agreement to participate in the patient's study
* Intellectual abilities compatible with the performance of cognitive or motor tasks

Exclusion Criteria:

* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (pregnant women, parturient women, mothers, etc.) who is breastfeeding, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure
* Patients in whom transient cessation of stimulation is not tolerated
* Subject in period of exclusion from another study
* Subject cannot be contacted in case of emergency
* Subject under administrative or judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pathologies included will be Parkinson's disease (PD), essential tremor, dystonia, and obsessive compulsive disorder (OCD).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Behavioral effect of DBS on confidence | by fall 2024
  Confidence in correct and incorrect responses will be compared on and off stimulation

SECONDARY OUTCOMES:
Effect of DBS on EEG markers of confidence | by fall 2024
  EEG correlates of confidence in correct and incorrect responses will be compared on and off stimulation

CONTACTS AND LOCATIONS:
Overall Officials: ELENA MORO, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: Yes
Experimental paradigms, anonymized behavioral and EEG data and analysis scripts will be made freely available on dedicated platforms (e.g zenodo)
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared upon publication of results, for an unlimited duration.